CLINICAL TRIAL: NCT01575405
Title: A Randomized, Double Blind Phase 1 Safety, Acceptability, and Pharmacokinetic Study Comparing Three Formulations of Tenofovir 1% Gel Administered Rectally to HIV-1 Seronegative Adults
Brief Title: A Study to Compare Three Different Formulations of Tenofovir 1% Gel When Administered Rectally
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ian McGowan (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); CONRAD (Other)
Responsible Party: Sponsor-Investigator, Ian McGowan, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CHARM-01; 5U19AI082637 (NIH)
Record Dates: First submitted 2012-02-29; First posted 2012-04-11 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Tenofovir; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rectal-specific formulation (RF) stage (Experimental): During this stage, participants will receive seven rectally-administered doses of the rectal-specific formulation (RF), with the first and last dose administered in clinic and five doses in between self-administered by a participant at home. Various specimens will be collected after administration of the last dose, including blood, vaginal and rectal fluids, and endoscopic biopsies. Blood and fluids will be additionally collected at 2hr, 4hr, and 24hr post-last-dose administration.
  Interventions: Drug: Rectal formulation (RF) of tenofovir 1% gel
- Vaginal formulation (VF) stage (Active Comparator): During this stage, only one exposure to the vaginal formulation (VF) will be administered (as the seventh dose in the stage), but it will be coupled with six preceding exposures to the Universal HEC Placebo Gel to balance it out against the other three stages in the study.
  First and last doses will be administered in clinic, and after the administration of the last dose, various specimens will be collected, including blood, vaginal and rectal fluid, and endoscopic biopsies. Additional blood and fluids will be collected at 2, 4, and 24 hours post seventh dose administration.
  Interventions: Drug: Vaginal formulations (original VF and reduced vaginal glycerin formulation RGVF) of tenofovir 1% gel; Drug: Universal HEC Placebo Gel Formulation
- Reduced Glycerin Vaginal Formulation (RGVF) stage (Active Comparator): During this stage, participants will receive seven rectally-administered doses of the reduced glycerin vaginal formulation (RGVF), with the first and last dose administered in clinic and five doses in between self-administered by a participant at home. Various specimens will be collected after administration of the last dose, including blood, vaginal and rectal fluids, and endoscopic biopsies. Blood and fluids will be additionally collected at 2hr, 4hr, and 24hr post-last-dose administration.
  Interventions: Drug: Vaginal formulations (original VF and reduced vaginal glycerin formulation RGVF) of tenofovir 1% gel

INTERVENTIONS:
Drug: Rectal formulation (RF) of tenofovir 1% gel — The RF is a translucent colorless viscous gel formulation containing 1% (w/w) of tenofovir (PMPA) formulated in purified water with EDTA, glycerin, methylparaben, propylparaben, carbopol, sodium carboxy methyl cellulose, and pH adjusted to 7. The RF is close to isoosmolar with an osmolality of 479 mOsmol/kg. Seven doses of this formulation will be used.
  Arms: Rectal-specific formulation (RF) stage
Drug: Vaginal formulations (original VF and reduced vaginal glycerin formulation RGVF) of tenofovir 1% gel — The original VF is a transparent, viscous gel formulation containing 1% (weight/weight) of tenofovir (PMPA, 9-[(R)-2-(phosphonomethoxy) propyl]adenine monohydrate), formulated in purified water with edetate disodium, citric acid, glycerin, methylparaben, propylparaben, hydroxyethylcellulose, and pH adjusted to 4-5. One dose of this formulation will be used, with 6 doses of the HEC placebo gel preceding it to balance out this study stage. The reduced glycerin formulation (RGVF) is a modification of the original VF - it has lower glycerin content than the VF and a significantly reduced osmolality (836 or 846 versus 3111 mOsmol/kg). Lowering the glycerin content lowered the viscosity, so the HEC concentration was increased by 10% (a change considered to be insignificant). The amount of parabens was increased by 10% each to improve the antimicrobial effectiveness. The RGVF formulation has since been modified to increase the viscosity. Seven doses of RGVF will be used in this study.
  Arms: Reduced Glycerin Vaginal Formulation (RGVF) stage; Vaginal formulation (VF) stage
Drug: Universal HEC Placebo Gel Formulation — The Universal HEC Placebo Gel contains hydroxyethylcellulose as the gelling agent, purified water, sodium chloride, sorbic acid and sodium hydroxide. The gel is isotonic and formulated at a pH of 4.4 to avoid disrupting the normal vaginal pH and has minimal buffering capacity to avoid the inactivation of sexually transmitted pathogens. Hydroxyethylcellulose is used to approximate the viscosity of microbicide gel candidates. Each pre-filled applicator will deliver approximately 4 mL of HEC placebo gel. Six doses of this gel will be used to balance out the VF stage of the study.
  Arms: Vaginal formulation (VF) stage

SUMMARY:
This is a double-blinded, randomized, safety, acceptability, pharmacokinetic, and ex vivo efficacy study of three rectally-applied tenofovir-based microbicide formulations. Approximately 18 total evaluable HIV-negative men and women (~9 per site) will be enrolled across two study sites: University of California at Los Angeles (UCLA) and Magee-Womens Research Institute (MWRI) at University of Pittsburgh.

Each participant will experience seven rectal exposures to the rectal-specific formulation (RF) and seven rectal exposures to the reduced glycerin vaginal formulation (RGVF) of tenofovir 1% gel, but only one exposure to the vaginal formulation (VF), which will be coupled with six preceding exposures to the Universal HEC Placebo Gel to balance out the VF study stage. Participant accrual will take approximately 6 months and each participant will be on study for approximately 3 months. The total duration of the study will be approximately 1 year.

The primary objectives of the study are safety, acceptability, and pharmacokinetics, specifically:

* To evaluate the safety of each tenofovir-based microbicide gel formulation when applied rectally
* To evaluate the acceptability of each tenofovir-based microbicide gel formulation when applied rectally
* To compare systemic and compartment pharmacokinetics among the three tenofovir-based microbicide gel formulations when applied rectally

Secondary objective of the study is to evaluate the mucosal immunotoxicity of each tenofovir-based microbicide gel formulation when applied rectally.

And the exploratory objective of the study is to assess the preliminary (ex vivo) efficacy of each tenofovir-based microbicide gel formulation using biopsy explants after each product is applied rectally.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ Age of 18 at screening
2. Willing and able to communicate in English
3. Willing and able to provide written informed consent to take part in the study
4. Willing and able to provide adequate locator information
5. Understands and agrees to local sexually transmitted infection (STI) reporting requirements
6. HIV-1 uninfected at screening according to the standard DAIDS algorithm in Appendix II
7. Must have been vaccinated for or have natural immunity to Hepatitis B, which will be verified by a positive Hepatitis B surface antibody (HBsAb) test at screening (Note: One re-screen will be allowed for individuals who are non immune to Hepatitis B but undergo vaccination.)
8. Availability to return for all study visits, barring unforeseen circumstances
9. Willing to abstain from RAI and practices involving insertion of anything in rectum (drug, enema, penis, or sex toy) for 72 hours before and 72 hours after each flexible sigmoidoscopy and study product exposure.
10. Must agree to use study provided condoms for the duration of the study
11. Must be in general good health
12. Must agree not to participate in other concurrent interventional and/or drug trials
13. Per participant report at screening, a history of consensual RAI at least once in the last three months.

    In addition to the criteria listed above, female participants must meet the following criteria:
14. Willing to abstain from insertion of anything into vagina (drug, douche, penis, or sex toy) other than the swabs/sponges for study related specimen collection for 24 hours before and after each study product exposure
15. Post-menopausal or using (or willing to use) an acceptable form of contraception (e.g., intrauterine device (IUD), hormonal contraception, surgical sterilization, or vasectomization of male partner). If the female participant has female partners only, the method of contraception will be noted as a barrier method in the study documentation. Temporary abstinence due to absence of partner(s) for the duration of the study will be acceptable.

Exclusion Criteria:

1. Abnormalities of the colorectal mucosa, or significant colorectal symptom(s), which in the opinion of the clinician represents a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids).
2. At screening: participant-reported symptoms and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current CDC guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include symptomatic bacterial vaginosis, symptomatic vaginal candidiasis, other vaginitis, trichomoniasis, Chlamydia (CT), gonorrhea (GC), syphilis, active HSV lesions, chancroid, pelvic inflammatory disease, genital sores or ulcers, cervicitis, or symptomatic genital warts requiring treatment. Note that an HSV-1 or HSV-2 seropositive diagnosis with no active lesions is allowed, since treatment is not required. (Note: In cases of non-anorectal GC/CT identified at screening, one re-screening 2 months after screening visit will be allowed.)
3. Per participant report and/or clinical or laboratory diagnosis, anorectal STI within six months prior to the Screening Visit
4. At screening:

   1. Hemoglobin < 10.0 g/dL
   2. Platelet count less than 100,000/mm3
   3. White blood cell count < 2,000 cells/mm3 or > 15,000 cells/mm3
   4. For females: calculated creatinine clearance less than 60 mL/min by the Cockcroft-Gault formula where creatinine clearance in mL/min (140- age in years) x (weight in kg) x (0.85 for female)/72 x (serum creatinine in mg/dL)
   5. For males: calculated creatinine clearance less than 60 mL/min by the Cockcroft-Gault formula where creatinine clearance in mL/min = (140 - age in years) x (weight in kg) x (1 for male)/72 x (serum creatinine in mg/dL)
   6. Serum creatinine > 1.3× the site laboratory upper limit of normal (ULN)
   7. Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 2.5× the site laboratory ULN
   8. +1 glucose or +1 protein on urinalysis (UA)
   9. History of bleeding problems (verified via prothrombin time (PT)/ International Normalized Ratio (INR) test)
   10. Positive for Hepatitis B surface antigen (HBsAg)
5. History of significant gastrointestinal bleeding in the opinion of the investigator
6. Known allergic reaction to methylparaben, propylparaben, sorbic acid, glycerin, glycerol, or tenofovir
7. Current known HIV-infected partner(s)
8. By participant report at enrollment, history of excessive daily alcohol use (as defined by the CDC as heavy drinking consisting of an average consumption of more than 2 drinks per day for men, and more than 1 drink per day for women), frequent binge drinking or illicit drug use that includes any injection drugs, methamphetamines (crystal meth), heroin, or cocaine including crack cocaine, within the past 12 months
9. Per participant report at screening, anticipated use and/or unwillingness to abstain from the following medications during the period of study participation:

   1. Heparin, including Lovenox®
   2. Warfarin
   3. Plavix® (clopidogrel bisulfate)
   4. Rectally administered medications (including over-the-counter products)
   5. Acyclovir, valacyclovir, famciclovir, and TDF
   6. >81 mg of aspirin per day AND unwillingness and/or inability to completely stop all use of aspirin or aspirin-containing medications for 3 days before and 3 days after the biopsy collection procedure
   7. Non-steroidal anti-inflammatory drugs (NSAIDS)
   8. Any other drugs that are associated with increased likelihood of bleeding following mucosal biopsy
10. By participant report at screening, use of systemic immunomodulatory medications, rectally administered medications, rectally administered products (including condoms) containing N-9, or any investigational products within the 4 weeks prior to the Enrollment/Baseline Evaluation Visit and throughout study participation
11. History of recurrent urticaria
12. Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease

    In addition to the criteria listed above, female participants will be excluded if they meet any of the following criteria:
13. Pregnant at the Enrollment/Baseline Visit
14. Breastfeeding at screening or intend to breastfeed during study participation per participant report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events and/or abnormal laboratory values Grade 2 or higher | Participants will be followed for the duration of study, an expected average of 12 weeks
  Grade 2 or higher clinical and laboratory adverse events as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 and Addenda 1 and 3 (Female Genital and Rectal Grading Tables for Use in Microbicide Studies) will be used to assess safety.
Proportion of participants reporting product characteristics as barriers in use | 24 hours post seventh dose administration of each study product
  We will calculate the proportion of participants who report product characteristics to be considered a barrier in use, operationalized as having a rating of lower than 3 on a 5-point Likert scale, in disliking or likelihood of future barrier in use. The phone interviews will be audio-taped, transcribed, and analyzed for content. In this process, we will be able to integrate the qualitative data to gain insights about the quantitative responses.
Area Under Curve (AUC) | 30 min, 2hr, 4hr, and 24hr post-dose at Visits 4, 5, 7, 8, 10, and 11
  Tenofovir concentrations will be measured via:
  * Plasma
  * PBMC (intracellular)
  * Rectal fluid
  * Vaginal fluid, in female participants
  * Rectal mucosal tissue homogenates
  * Rectal MMC
  Tenofovir diphosphate concentrations will be measured via:
  * PBMC
  * Rectal mucosal tissue homogenates
  * Rectal MMC

SECONDARY OUTCOMES:
Changes in rectal microflora | 30 min before first dose and 24 hr after seventh dose of each study gel
  Microflora measures will be graded on a 0 to 4 ordinal scale and recorded at baseline and post-exposure. Depending on the empirical distributions across the points in this scale, statistical procedures will either involve analysis of the actual pre-post differences (ordinal) or dichotomized versions of the pre and post scores (binary).
Changes in cytokine levels in rectal secretions | 30 min before first dose, 30 min before seventh dose, and 24 hr after seventh dose of each study gel
  Comparisons will be used to examine whether (i) there is an overall change in cytokine levels before/after (24 hours) each product exposure and (ii) whether the study products differ significantly from each other in pre-post change.
Changes in rectal histology | 30 min post seventh dose of each study gel
  Examination of two point (normal versus abnormal) or three point (normal, slightly abnormal, abnormal) scales will be undertaken. As above, comparisons will be used to examine whether (i) there is an overall change in histology scores before/after (24 hours) each product exposure and (ii) whether the study products differ significantly from each other in pre-post change.
Changes in rectal tissue CD4 cell phenotype | 30 min post seventh dose of each study gel
  comparisons will be used to examine whether (i) there is an overall change in cell populations before/after (24 hours) each product exposure and (ii) whether the study products differ significantly from each other in pre-post change.
Changes in intestinal mucosal cytokine mRNA levels | 30 min post administration of seventh dose each study gel
  mRNA levels will be used to evaluate stability (intra-subject correlations) and clinically meaningful differences between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ian McGowan, MD, PhD, FRCP, Study Chair — Magee-Women's Research Institute
Locations (2):
- United States (2):
  - UCLA Center for Prevention Research, Los Angeles, California
  - Magee/University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Mcgowan I, Cranston RD, Duffill K, Siegel A, Engstrom JC, Nikiforov A, Jacobson C, Rehman KK, Elliott J, Khanukhova E, Abebe K, Mauck C, Spiegel HM, Dezzutti CS, Rohan LC, Marzinke MA, Hiruy H, Hendrix CW, Richardson-Harman N, Anton PA. A Phase 1 Randomized, Open Label, Rectal Safety, Acceptability, Pharmacokinetic, and Pharmacodynamic Study of Three Formulations of Tenofovir 1% Gel (the CHARM-01 Study). PLoS One. 2015 May 5;10(5):e0125363. doi: 10.1371/journal.pone.0125363. eCollection 2015. PMID 25942472